CLINICAL TRIAL: NCT05109728
Title: A Phase Ib Dose Finding Study Assessing Safety and Activity of [177Lu]Lu-DOTA-TATE in Newly Diagnosed Glioblastoma in Combination With Radiotherapy With or Without Temozolomide and in Recurrent Glioblastoma as Single Agent
Brief Title: A Dose Finding Study of [177Lu]Lu-DOTA-TATE in Newly Diagnosed Glioblastoma in Combination With Standard of Care and in Recurrent Glioblastoma as a Single Agent.
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAAA601A52101; 2021-003672-14 (EudraCT Number)
Record Dates: First submitted 2021-10-27; First posted 2021-11-05 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; GBM; Radioligand Therapy; RLT; [177Lu]Lu-DOTA-TATE; Temozolomide; O-6-methylguanine-DNA methyltransferase; MGMT
MeSH Terms: conditions — Glioblastoma | interventions — lutetium Lu 177 dotatate; Temozolomide; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 - Newly diagnosed GB (Experimental): Participants with newly diagnosed glioblastoma will receive [177Lu]Lu-DOTA-TATE every 4 weeks +/- 2 days, starting 7 to 10 days prior to initiation of Radiotherapy (RT) and Temozolomide (TMZ)
  Interventions: Drug: [177Lu]Lu-DOTA-TATE; Drug: [68Ga]Ga-DOTA-TATE; Other: Temozolomide; Other: Radiotherapy
- Group 3 - Recurrent GB (Experimental): Participants with recurrent glioblastoma will receive [177Lu]Lu-DOTA-TATE as single agent therapy every 3 weeks +/- 2 days
  Interventions: Drug: [177Lu]Lu-DOTA-TATE; Drug: [68Ga]Ga-DOTA-TATE

INTERVENTIONS:
Drug: [177Lu]Lu-DOTA-TATE — Group 1: [177Lu]Lu-DOTA-TATE, dose level 0 (150mCi) administered every 4 weeks. Three provisional dose levels (Dose level +2: 250 mCi; Dose level +1: 200 mCi; Dose level -1: 100 mCi) will be assessed.
  Group 3: [177Lu]Lu-DOTA-TATE, dose level 0 (150mCi) administered every 3 weeks. Three provisional dose levels (Dose level +2: 250 mCi; Dose level +1: 200 mCi; Dose level -1: 100 mCi) will be assessed.
  Other Names: Lutathera; Lutetium (177Lu)oxodotreotide; Lutetium Lu 177dotatate
Drug: [68Ga]Ga-DOTA-TATE — 2 MBq/kg of body weight (0.054 mCi/kg), with a minimum dose of 100 MBq (2.7 mCi) and maximum dose of 200 MBq (5.4 mCi)
Other: Temozolomide — Concomitant Phase: Temozolomide 75mg/m2/d p.o until last day of EBRT.
  Maintenance Phase: Temozolomide p.o 150 mg/m2/d during cycle 1 then 200 mg/m2/d for the following cycles if tolerated well in Cycle 1. 6 cycles total (1 cycle = every 28 days)
  Arms: Group 1 - Newly diagnosed GB
Other: Radiotherapy — 2 Gy/day, 5 days per week followed by 2 days of rest, for 6 consecutive weeks
  Arms: Group 1 - Newly diagnosed GB

SUMMARY:
A Dose Finding Study of [177Lu]Lu-DOTA-TATE in Newly Diagnosed Glioblastoma in Combination with Standard of Care and in Recurrent Glioblastoma as a Single Agent

DETAILED DESCRIPTION:
The study for each participant consists of a Screening period, a Treatment period and a 12-month Follow-up period.

During the screening period of up to 6 weeks before starting GBM treatment, each participant will be assessed for somatostatin receptor (SSTR) expression by [68Ga]Ga-DOTA-TATE imaging PET/scan.

Eligible participants with newly diagnosed glioblastoma will be assigned to Group 1 :

• Participants in Group 1 (concomitant radiotherapy + temozolomide and temozolomide maintenance) will receive treatment with [177Lu]Lu-DOTA-TATE every 4 weeks +/- 2 days, up to 6 administrations. Radiotherapy and temozolomide will be administered 7 to 10 days after the first administration of [177Lu]Lu-DOTA-TATE. Temozolomide will be administered orally at a dose of 75 mg/m2/day during the concomitant period, concurrently with radiotherapy. Radiotherapy will be delivered at a dose of 2 Gray (Gy)/day, 5 days per week followed by 2 days of rest, for 6 consecutive weeks with a total dose of 60 Gy (without interruption). During the maintenance period, there is an intra-patient dose escalation in temozolomide treatment. The dosage of temozolomide is 150 mg/m2 in Cycle 1 of maintenance period, and then to 200 mg/m2 in Cycle 2 and beyond in the maintenance period, if 150 mg/m2 temozolomide treatment is well tolerated in Cycle 1.

Eligible participants with recurrent glioblastoma will be assigned to Group 3 and will receive [177Lu]Lu-DOTA-TATE as single agent treatment every 3 weeks +/- 2 days.

An infusion of sterile 2.5% Lysine - Arginine amino acid (AA) solution will be co-administered with each [177Lu]Lu-DOTA-TATE dose for renal protection.

ELIGIBILITY:
Key Inclusion Criteria:

Common Criteria:

* Participant is >= 18 years on the day of signing informed consent form
* Histologically confirmed glioblastoma
* Adequate bone marrow, organ function and electrolyte values

Newly diagnosed glioblastoma (Group 1):

* Presence of Gadolinium enhancing tumor in pre-surgery magnetic resonance imaging (MRI)
* Karnofsky Performance Score (KPS) >= 70 %

Recurrent glioblastoma (Group 3 dose Escalation only):

• Participant has experienced first or second recurrence of their glioblastoma, after standard or experimental therapy that includes prior EBRT

Recurrent glioblastoma (Group 3 dose escalation and expansion):

* Evidence of recurrent disease demonstrated by disease progression using modified Response Assessment in Neuro-Oncology (mRANO) criteria
* KPS >= 60 %
* [68Ga]Ga-DOTA-TATE uptake by positron emission tomography/computed tomography (PET/CT) or PET/MRI at the tumor region
* Presence of Gadolinium enhancement in the tumor region in MRI at the time of diagnosis of tumor recurrence
* A second surgery for glioblastoma is allowed provided that the following criteria are met:

  1. Residual and measurable disease post-surgery is not required but surgery must have confirmed the diagnosis of recurrence
  2. Surgery completed at least 2 weeks prior to study treatment initiation, with post-surgery recovery without any complications related to surgical procedure

     Recurrent glioblastoma (Group 3 Dose Expansion only):
* Patients experiencing first recurrence of their glioblastoma, after standard or experimental therapy that includes prior EBRT

Key Exclusion Criteria:

Common Criteria:

* Participant is receiving additional, concurrent, active therapy for glioblastoma outside of the trial
* Extensive leptomeningeal disease
* History of another active malignancy in the previous 3 years prior to study entry
* Prior administration of a radiopharmaceutical unless 10 or more effective half-lives have elapsed before injection of [68Ga]Ga-DOTA-TATE or [177Lu]Lu-DOTA-TATE

Newly diagnosed glioblastoma (Group 1):

• Any prior treatment for glioma of any grade

Recurrent glioblastoma (Group 3 dose escalation and expansion):

* Early disease progression prior to 3 months from the completion of radiotherapy
* Previous treatment with bevacizumab for the treatment of glioblastoma with therapeutic intent, or with bevacizumab as supportive therapy (e.g. edema reduction) within 60 days of initiation of study treatment

Recurrent glioblastoma (Group 3 dose escalation only):

• More than 2 prior lines for systemic therapy

Recurrent glioblastoma (Group 3 dose expansion only):

• More than 1 prior line for systemic therapy

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-05-10 (Actual); Primary Completion 2026-06-05 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Group 1: Frequency of dose limiting toxicities (DLTs) | 49 to 52 days starting from first administration of [177Lu]Lu-DOTA-TATE
  A dose-limiting toxicity (DLT) is defined as an AE or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that meets any of the criteria defining dose-limiting toxicities and with an onset during the DLT observation period specified for the group.
  • Group 1: DLT observation period of 49 to 52 days starting from the first administration of [177Lu]Lu-DOTA-TATE (Day 1) and ending with the completion of concomitant RT and TMZ. The 49 to 52 days observation period is depending on the start day of concomitant RT and TMZ (i.e. 7-10 days post first [177Lu]Lu-DOTA-TATE dose). If the concomitant RT and TMZ is delayed for any reason, the DLT observation period will last until the completion of the concomitant treatment. If RT or TMZ is delayed, the DLT observation period will last until the last administered dose, whichever occurs later.
Group 3: Frequency of dose limiting toxicities (DLTs) | 42 days starting from first administration of [177Lu]Lu-DOTA-TATE
  A dose-limiting toxicity (DLT) is defined as an AE or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that meets any of the criteria defining dose-limiting toxicities and with an onset during the DLT observation period specified for the group.
  • Group 3: DLT observation period of 42 days starting from the first administration of [177Lu]Lu-DOTA-TATE (Day 1) i.e. accounting for 2 cycles of Lu]Lu-DOTA-TATE.

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs), serious AEs (SAEs) of [177Lu]Lu-DOTA-TATE | Up to approximately 2 years (estimated final OS analysis) from date of first study treatment
  The distribution of adverse events of [177Lu]Lu-DOTA-TATE will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
  During the follow up period, all AEs and lab abnormalities will be collected within 8 weeks after the last dose of study treatment. For participants with study drug related AEs, they will be followed until resolution or until the End of Study, whichever occurs first. Apart from that, only survival information, SAEs, that are considered related to study drug by the Investigator, and AEs of secondary hematological malignancies will be collected until the end of follow up period every 8 weeks.
Incidence and severity of Adverse Events (AEs) and serious Adverse Events (SAEs) within 48 hours after [68Ga]Ga-DOTA-TATE infusion | up to 48 hours following the start of [68Ga]Ga-DOTA-TATE administration
  The distribution of adverse events of [68Ga]Ga-DOTA-TATE will be done via the analysis of frequencies for treatment emergent Adverse Event (TEAEs), Serious Adverse Event (TESAEs) and Deaths due to AEs, through the monitoring of relevant clinical and laboratory safety parameters.
Overall Objective Status as per modified Response Assessment in Neuro-Oncology (mRANO) criteria | Up to approximately 2 years (estimated final OS analysis) from date of first study treatment
  According to modified RANO, the objective overall status combines the radiographic response on target lesions, new disease, neurological status and use of steroids and the result is reported as confirmed or preliminary CR, confirmed or preliminary PR, stable disease, confirmed or preliminary disease progression. The best objective overall status achieved during the study will be summarized using frequency and percentage. The rate of confirmed complete or partial response will be summarized using point estimate and 2-sided exact binomial 95% confidence interval (Clopper-Pearson) and presented by dose level within each group.
Progression-Free Survival (PFS) | From date of randomization until date of progression or date of death from any cause, whichever come first, assessed for up to 2 years (estimated final OS analysis)
  Progression-Free Survival (PFS) is defined as the time from the date of first dose to the date of confirmed progression according to modified RANO or death due to any cause. If no PFS event is observed, PFS will be censored at the date of the last adequate tumor assessment prior to data cut-off date and start of new anti neoplastic therapy, whichever comes first. PFS will be analyzed in the FAS population and results will be presented for each dose level within each group. The PFS distribution will be estimated using the Kaplan-Meier method.
Overall Survival (OS) | Up to approximately 2 years (estimated final OS analysis) from date of first study treatment
  Overall Survival (OS) is defined as the time from date of first dose to date of death due to any cause. If a participant is not known to have died, then OS will be censored at the latest date the participant was known to be alive (on or before the cut-off date). OS will be analyzed in the FAS population and results will be presented for each dose level within each group. The OS distribution will be estimated using the Kaplan-Meier method.
Group 1: Time activity curves (TACs) | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Time activity curves (TACs), describing percentage (%) of the activity injected vs time in blood, organs and tumor lesions
Group 1: Absorbed radiation doses of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Absorbed radiation doses of [177Lu]Lu-DOTA-TATE in organs and tumor lesions will be summarized with descriptive statistics.
Group 1: Concentration of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Blood samples for radioactivity measurement will be collected before the start of [177Lu]Lu-DOTA-TATE infusion, at the end of [177Lu]Lu-DOTA-TATE infusion, then at 2 h, 6 h, 24 h, 48 h and 168 h after the end of [177Lu]Lu-DOTA-TATE infusion for participants undergoing dosimetry. Blood samples will be drawn in heparinized tubes. Radioactivity measurements on blood will be performed locally on site, using a gamma-counter.
Group 1: Observed maximum plasma concentration (Cmax) of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Cmax will be listed and summarized using descriptive statistics.
Groups 1: Time of maximum observed drug concentration occurrence (Tmax) of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Tmax will be listed and summarized using descriptive statistics.
Group 1: Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity-based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. AUClast will be listed and summarized using descriptive statistics.
Group 1: Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. AUCinf will be listed and summarized using descriptive statistics.
Group 1: Total systemic clearance for intravenous administration (CL) of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. CL will be listed and summarized using descriptive statistics.
Group 1: Volume of distribution during the terminal phase following intravenous elimination (Vz) of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Vz will be listed and summarized using descriptive statistics.
Group 1: Terminal elimination half-life (T^1/2) of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. The half-life will be listed and summarized using descriptive statistics.
Group 1: Terminal-Phase Disposition Rate Constant (λz) of [177Lu]Lu-DOTA-TATE | Week 5 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 5 Day 2 (24 hours post-dose), Week 5 Day 3 (48 hours post-dose), Week 5 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Terminal-Phase Disposition Rate Constant will be listed and summarized using descriptive statistics.
Group 3: Time activity curves (TACs) | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Time activity curves (TACs), describing percentage (%) of the activity injected vs time in blood, organs and tumor lesions
Group 3: Absorbed radiation doses of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Absorbed radiation doses of [177Lu]Lu-DOTA-TATE in organs and tumor lesions will be summarized with descriptive statistics.
Group 3: Concentration of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Blood samples for radioactivity measurement will be collected before the start of [177Lu]Lu-DOTA-TATE infusion, at the end of [177Lu]Lu-DOTA-TATE infusion, then at 2 h, 6 h, 24 h, 48 h and 168 h after the end of [177Lu]Lu-DOTA-TATE infusion for participants undergoing dosimetry. Blood samples will be drawn in heparinized tubes. Radioactivity measurements on blood will be performed locally on site, using a gamma-counter.
Group 3: Observed maximum plasma concentration (Cmax) of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Cmax will be listed and summarized using descriptive statistics.
Group 3: Time of maximum observed drug concentration occurrence (Tmax) of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Tmax will be listed and summarized using descriptive statistics.
Group 3: Area under the serum concentration-time curve from time zero to the time of last quantifiable concentration (AUClast) of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity-based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. AUClast will be listed and summarized using descriptive statistics.
Group 3: Area under the concentration-time curve from time zero (pre-dose) extrapolated to infinite time (AUCinf) of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. AUCinf will be listed and summarized using descriptive statistics.
Group 3: Total systemic clearance for intravenous administration (CL) of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. CL will be listed and summarized using descriptive statistics.
Group 3: Volume of distribution during the terminal phase following intravenous elimination (Vz) of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Vz will be listed and summarized using descriptive statistics.
Group 3: Terminal elimination half-life (T^1/2) of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. The half-life will be listed and summarized using descriptive statistics.
Group 3: Terminal-Phase Disposition Rate Constant (λz) of [177Lu]Lu-DOTA-TATE | Week 4 Day 1 (pre-dose, before the end of infusion, 2 hours post-dose, 6 hours post-dose), Week 4 Day 2 (24 hours post-dose), Week 4 Day 3 (48 hours post-dose), Week 4 Day 8 (168 hours post-dose)
  Venous whole blood samples will be collected and analysed for radioactivity. Radioactivity based concentration units will be converted to mass-based concentration units using the specific activity of the dose at the time of manufacture (MBq/µg). Pharmacokinetics characterization will be performed on mass-based concentrations. Terminal-Phase Disposition Rate Constant will be listed and summarized using descriptive statistics.
Quantification of [177Lu]Lu-DOTA-TATE excreted from the body in urine | From the start of [177Lu]Lu-DOTA-TATE infusion until the first whole body planar imaging
  All excreted urine from the start of [177Lu]Lu-DOTA-TATE infusion until the first whole body planar imaging will be collected, its volume measured and the radioactivity concentration kilobecquerel per milliliter (kBq/mL) determined in order to calculate the total radioactivity excreted from the body from the start of [177Lu]Lu-DOTA-TATE infusion to the time of the first scan. If no urine is excreted from the start of [177Lu]Lu-DOTA-TATE infusion until the first whole body planar imaging, no urine dosimetry is necessary.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (13):
- United States (5):
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Col Uni Med Center New York Presby, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - MD Anderson Cancer Center Uni of Te, Houston, Texas
  - University of Wisconsin School of Medicine and Public Health, Madison, Wisconsin
- France (2):
  - Novartis Investigative Site, Bron
  - Novartis Investigative Site, Marseille
- Novartis Investigative Site, Porto, Portugal
- Spain (3):
  - Novartis Investigative Site, Granada, Andalusia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid
- Switzerland (2):
  - Novartis Investigative Site, Lausanne
  - Novartis Investigative Site, Zurich

IPD SHARING:
Plan to Share IPD: No